CLINICAL TRIAL: NCT02167126
Title: Kinesio Taping Effects on Knee Extension Force Among Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Franca (Other)
Responsible Party: Principal Investigator, Paulo Roberto Veiga Quemelo, Paulo Quemelo, University of Franca
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UFranca02
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Kinesio Taping Effects on Knee Extension Force
Keywords: Athletic Performance;; Muscle Strength;; Isometric Contraction;; Kinesio Taping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio Taping (Experimental): Kinesio Taping was applied as experimental group.
  Interventions: Device: Kinesio Taping; Device: Placebo Tape
- Micropore (Placebo Comparator): Micropore Tape was used as placebo tape
  Interventions: Device: Kinesio Taping; Device: Placebo Tape

INTERVENTIONS:
Device: Kinesio Taping — using the "V" technique, the knee was positioned at 45º of flexion, the origin of both tapes was located 10 cm below the anterior-superior iliac spine with one tape going laterally and one medially to the rectus femoris muscle belly, passing around the patella and finishing on the tibial tuberosity.
Device: Placebo Tape — Micropore tape was applied using the "V" technique, the knee was positioned at 45º of flexion, the origin of both tapes was located 10 cm below the anterior-superior iliac spine with one tape going laterally and one medially to the rectus femoris muscle belly, but because it is not elastic, the knee joint was not crossed and the end points were the medial and lateral aspects of the patella.

SUMMARY:
Kinesio Taping (KT) is used often, but there is little scientific information on its effect. The aim of this study was to evaluate the effects of KT on knee extension force among soccer players. KT (K-Tape®) and Micropore (3M®) were applied on the right and left thighs of 34 professional soccer players (20 males and 14 females). Half of the participants had KT applied to the left and half to the right thigh. The subjects performed two maximal isometric voluntary contractions of the quadriceps pre, immediately post, and 24 hours after tape application. Isometric knee extension force was measured using a load cell and the following variables were assessed: peak force, time to peak force, rate of force development until peak force, time to peak rate of force development and 200 ms pulse. There were no statistically significant differences between KT and Micropore conditions or among testing sections (pre, post, and 24h after). Therefore, taping (independently of the type of tape used or time since application) did not affect the force-related measures assessed during maximal isometric voluntary knee extension trials performed by healthy professional athletes.

DETAILED DESCRIPTION:
Kinesio taping was applied on the skin over the rectus femoris muscle on one limb and 3M Micropore® (placebo tape) was applied on the contralateral limb. Different tapes were used to evaluate if tape type would affect the findings. The side of application of the different tapes was randomized among the participants. Half of the participants (n = 17) had KT applied to the left thigh and the other half to the right thigh (n = 17). KT was applied using the "V" technique, the knee was positioned at 45º of flexion, the origin of both tapes was located 10 cm below the anterior-superior iliac spine with one tape going laterally and one medially to the rectus femoris muscle belly, passing around the patella and finishing on the tibial tuberosity. The same technique was used for the Micropore tape on the contralateral limb, but because it is not elastic, the knee joint was not crossed and the end points were the medial and lateral aspects of the patella. The mean force values were calculated for each condition (pre, post and 24 hours after tape application). The isometric knee extension force was collected using a load cell (EMG System do Brasil Ltda. ®) with a measuring range from 0 to 200 kg at 1000 Hz, filtered with a low pass filter type Butterworth 4th order and cut-off frequency of 15 Hz, obtained through residual analysis.

ELIGIBILITY:
Inclusion Criteria:

* To participate the athletes had to be at least 18 years old and not have lower limb injuries at the time of testing

Exclusion Criteria:

* Younger than 18 years old

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Knee extension force | 24 hours
  To evaluate the effects of Kinesio Taping on knee extension force among soccer players. The participants performed two five-second maximal isometric voluntary knee extension trials during three testing sections: pre, immediately post, and 24 hours after application of the tapes.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RV Quemelo, PhD, Principal Investigator — Universidade de Franca
Locations (1):
- University of Franca, Franca, São Paulo, Brazil

REFERENCES:
- [Result] Hsu YH, Chen WY, Lin HC, Wang WT, Shih YF. The effects of taping on scapular kinematics and muscle performance in baseball players with shoulder impingement syndrome. J Electromyogr Kinesiol. 2009 Dec;19(6):1092-9. doi: 10.1016/j.jelekin.2008.11.003. Epub 2009 Jan 14. PMID 19147374
- [Derived] Serra MV, Vieira ER, Brunt D, Goethel MF, Goncalves M, Quemelo PR. Kinesio Taping effects on knee extension force among soccer players. Braz J Phys Ther. 2015 Mar-Apr;19(2):152-8. doi: 10.1590/bjpt-rbf.2014.0075. Epub 2015 Mar 13. PMID 25789557